CLINICAL TRIAL: NCT05831722
Title: Changes in the Upper Airway Volume After Rapid Maxillary Expansion in Adults Using Pure Skeletal Anchorage
Status: Completed | Type: Observational
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, JAVIER MONTERO, Director, University of Salamanca
Other Study IDs: USAL 2023-AZM
Record Dates: First submitted 2023-04-11; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Orthodontic Appliance Complication; Dental Malocclusion; Bone Anchored Rapid Maxillary Expansion; Maxillary Hypoplasia; BAME
MeSH Terms: conditions — Malocclusion; Retrognathia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Rapid Maxillary Expansion — Rapid Maxillary Expansion consists in the mid palatal suture opening through temporary anchorage mini implants placed in the palatal area.

SUMMARY:
The objective of this study is to evaluate the effect of bone-anchored rapid maxillary expansion (RME) in the volume of the right maxillary sinus, left maxillary sinus and nasal and maxillary sinus airway complex, through bone anchored maxillary expansion devices (BAME); in addition, the influence of gender and age in the volume changes will be also analyzed. Material and method: 18 patients between undergone RME treatment with a jackscrew based on 4 miniscrews which will be placed in the palate on both sides of the midpalatal suture. Cone-beam computed tomography (CBCT) scans will be taken before and after suture palatine expansion and datasets will be uploaded into therapeutic digital planning software to measure the volume (mm3) of the right maxillary sinus, left maxillary sinus (mm3) and nasal and maxillary sinus airway complex (mm3). The airway volumes will be isolated after selecting the anatomical area in the axial, coronal and sagittal space plane and ensuring the air density measurement by reference points placement inside the selected area. Statistical analysis between preoperative and postoperative measurements will be performed using the statistical analysis of the t-test.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* no history of systemic conditions that could interfere in bone metabolism and in the surgical process of orthodontic mini-implant placement
* radiographic imaging (CBCT KAVO OP3D Pro FOV 13X15cm) of maxillary discrepancy of more than 3mm compared with the ideal dimensions according to their mandible

Exclusion Criteria:

* Age more than 31 years old
* Systematic conditions that interfere in bone metabolism

Ages: 19 Years to 31 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: dental clinic patients
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
The paired t-test analysis will show any statistically significant differences between the preoperative and postoperative volumes of the nasal and maxillary sinus airway complex | 2 months after bone anchored maxillary expansion is completed

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Clinica Odontológica de la Universidad de Salamanca, Salamanca
  - Javier Montero, Salamanca
  - University of Salamanca, Salamanca